CLINICAL TRIAL: NCT04197648
Title: The Effect of Exercise on Thoracic Aortic Aneurysm and Blood Pressure Control.
Brief Title: Effects of Exercise on Thoracic Aneurysms
Acronym: EXTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Paul Poirier, Cardiologist, Laval University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-4350
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Intervention Model Description: Just before the intervention and baseline evaluation, each subject will be randomized either in the exercise or the control group.
  Experimental group (exercise): 12 week supervised exercise program. Control group: Daily life activities
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Exercise: 12 week, supervised exercise program. 3x/week.
  Interventions: Device: Exercise group
- Control goup (No Intervention): No exercise program. Continuation of the daily life activities. Consultation with a kinesiologist at baseline, 3 months and 6 months for advice on physical activities and lifestyle habits.

INTERVENTIONS:
Device: Exercise group — 24 week supervised exercise program (strength and cardiovascular program).
  Arms: Exercise group

SUMMARY:
Thoracic aneurysm incidence is estimated to 4.5 cases per 100 000. The manifestation as well as natural history of thoracic aneurysm depend on many factors such as its localisation, its diameter, presence of collagen disease and family history. For the ascendant aortic aneurysm, it is often linked to a degeneration of the media arterial layer of the arterial wall. The media degeneration is cause by the degeneration of the elastic fibres, which lead to a weakening of the arterial wall accompanied with dilation. This process is often due to age and is accelerated by high blood pressure. Amongst the numerous factors causing the aneurysm, the investigators find: hypertension, aortic bicuspid valve, smoking, atherosclerosis, trauma and genetic predisposition. The average growth rate of thoracic aneurysm is 0.1-0.2 cm/year. The risk of rupture is associated to the size of the aneurysm as well as patient's symptoms. The ruptures and dissections rates are accounted for 2-3/year for thoracic aneurysm between 5.5-6.0 cm in diameter. The patients are often limited in their daily life activities considering their concern and risk of rupture and/or dissect. The effects of exercise on the progression of the aneurysm dilation in patients with thoracic ascendant aortic aneurysm are unknown. It is well known that high blood pressure is a risk factor for rupture of the aortic aneurysm. Many studies have demonstrated the benefits of physical exercise regarding the lowering impact of blood pressure in a cardiac hypertensive population.

At 3 and 6 months of the intervention, the subjects in the exercise group will have: 1) a lowered blood pressure at rest and during exercise, 2) maintenance/ improvement of muscle strength, 3) improvement of aerobic exercise capacity (VO2max), and 4) aortic dilation that remained stable or comparable to the control group.

The research objective is to measure and compare to a control group, the effects of an exercise program on the following parameters: blood pressure response at rest and during exercise, as well as the VO2max at 3 and 6 months time of the intervention.

This randomised and prospective study will take place at the " Institut Universitaire de Cardiologie et de Pneumologie du Québec (IUCPQ) " and will include patients who have a non-surgical ascendant thoracic aortic aneurysm (ATAA). The selected subjects will be randomised into two groups: 1) exercise group (n=15), and 2) control group (n=15). Both groups will be met prior to the intervention (baseline) and at 3 and 6 months time of the intervention, and measures described below will be recorded.

DETAILED DESCRIPTION:
To this day, the impact and influence of physical activity in this population has been reported in very few studies, and all have been led in a population with abdominal aorta aneurysm (AAA). These studies conclude that patients should avoid lifting heavy loads as well as performing isometric muscular exercises since these maneuvers increase significantly intra-thoracic pressure as well as blood pressure. As for aerobic exercise, it is recommended that all patient wanting to participate in high intensity activities must perform a cardiopulmonary exercise test (VO2max) to ensure that the systolic blood pressure does no exceed 180 mmHg.

This study will enable us to know the effects of a moderate to high intensity exercise program (80% of anaerobic threshold) on blood pressure response in this population. This will also allow the quantification and qualification of the blood pressure changes following an exercise program as well as the safeness of such an intervention.

Anthropometric measures will be taken for both groups before, at 3 months and 6 months intervention. Firstly, the subjects will be measured using a stadiometer scaled in cm. Then, they will be weighed using a bio-impedance scale of the type InBody (InBody 520, Body Composition Analyzer) in order to measure body composition. The mass values and height will be used to calculate the body mass index (BMI). Finally, waist circumference will be measured directly on the abdomen on the level of the iliac crest using a measuring tape scaled in cm. Waist circumference will be used to assess indirectly abdominal obesity.

In order to measure blood pressure variations and the hypotensive effect of exercise, a 24-hour ambulatory blood pressure monitoring (ABPM) in both groups will be performed at baseline, at 3 months and at 6 months intervention. In the exercise group, the ABPM will also be performed on a consecutive first training session. The measure will be performed over a period of 24 hours. The measures will be taken every 30 minutes during the day and every hour during the night.

A cardiopulmonary exercise test will be performed before, at 3 months and at 6 months intervention, in order to asses the maximum aerobic capacity (VO2max) of the subjects in both groups. This test will take place on an ergometer cycle with electromagnetic brakes (Lode Recumbent, Groningen, Nederland) which allows to determine the work (watts) independently of the rpm. Subjects will breathe in a mouthpiece related to a gas analyser (MedGraphics, St-Paul, MN). Furthermore, a 12 derivation electrocardiogram (Cardioperfect Welch-Allyn, Skaneateles Falls, NY) measuring cardiac activity and an oximeter (N-395 Nellcor, Boulder, CO) measuring the blood oxygen saturation will be installed on the subject for the entire duration of the test. Finally, every two minutes during the test, blood pressure measure will be taken followed by the effort perception based on the modified Borg scale. This test is administered by a certified Clinical Exercise Specialist from the American College of Sport Medicine (ACSM) and supervised by a physician.

A strength evaluation will be performed for both groups before, 3 months and at 6 months intervention. In order to obtain a specific and reliable exercise prescription for each subject, the 1 maximal repetition (MR) will be estimated using linear equations <10 MR since it is not recommended to asses 1 MR in this population due to the high blood pressure that this type of evaluation generates.

Handgrip strength will be measured. In a standing position, the patient will perform a maximum muscle contraction of the hand (hand dynamometer). This test will be performed with the right and left hand alternately. Strength evaluation, including the preparation and explanations, will last approximately 45 minutes.

In order to note the energy expense of each participant in both groups, a wireless portable monitor SenseWearPro2 (SWA; Body Media, Pittsburgh, USA) will be used. This monitor is an armband that subjects will use at baseline, at 3 months and 6 months. It will be worn during 3 consecutive days, 2 weekdays and 1 day during the weekend. The subjects will wear the armband as soon as they wake up in the morning and will remove it at bedtime.

A CT scan will be performed prior to the study (inclusion criteria; recent CT scan < 6 months), and at the end of the intervention, at 6 months. These CT scans are clinically required for follow up of the aneurysm dilation measure post intervention.

Subjects randomized in the exercise group will follow a 24-week structured supervised exercise program at the "Pavillon de Prévention des Maladies Cardiaques (PPMC) ". Each subject will have a personalized program. The goal is to perform this program 3x/week, and each session will last approximately 60 minutes: 40 minutes high intensity intervals training on cycle ergometer and 20 minutes strength training (2-3 sets, 10-15 repetitions). If needed, every week, the kinesiologist will adjust each participant's exercise program accordingly. The kinesiologist will be certified clinical exercise specialist from the ACSM.

During every session, blood pressure will be monitored at rest, following 5 minutes seated, before and after the session. Blood pressure will be taken during the high intensity interval and one during the low intensity interval. Heart rate will also be monitored during the intervals in order to calculate the double product (HR x SBP).

Subjects in the control group will have a consultation at 3 and 6 months time of the intervention with the kinesiologist. The consultation will last 1 hour. They will be given general advice regarding physical activity as well as healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Have an interest in participating in a supervised exercise training program
* Aortic diameter between 3,5 and 5 cm

Exclusion Criteria

* Glomerular filtration rate below 30 mL/min/1.73m²
* Aortic diameter greater than or equal to 5.1 cm
* Progression of aortic diameter greater than or equal to 0.5 cm per year
* Allergy to iodine
* Aortic valve bicuspidy
* History of aortic surgery or cardiac surgery
* Presence of an aortic dissection, penetrating aortic ulcer, or intra-mural hematoma of the aorta
* Presence of Marfan syndrome or other genetic and/or congenital disease explaining the thoracic aortic aneurysm
* History of stroke
* Presence of peripheral artery disease
* History and/or presence of aortitis
* Known diagnosis of temporal arteritis or rheumatoid arthritis
* Presence of a pacemaker
* Major cognitive limitation that may affect adherence to visits
* Musculoskeletal limitation that restricts participation in the training program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Aneurysm diameter | At 3 months of intervention
  Aneurysm dilation diameter is stable or comparable to control group

CONTACTS AND LOCATIONS:
Overall Officials: Paul Poirier, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Not yet approve by our ERB. If we want/plan to share individual participant data, we need to obtain approval from our ERB.

REFERENCES:
- [Background] Isselbacher EM. Thoracic and abdominal aortic aneurysms. Circulation. 2005 Feb 15;111(6):816-28. doi: 10.1161/01.CIR.0000154569.08857.7A. No abstract available. PMID 15710776
- [Background] Carvalho RS, Pires CM, Junqueira GC, Freitas D, Marchi-Alves LM. Hypotensive response magnitude and duration in hypertensives: continuous and interval exercise. Arq Bras Cardiol. 2015 Mar;104(3):234-41. doi: 10.5935/abc.20140193. Epub 2014 Dec 16. PMID 25517389
- [Background] Reynolds JM, Gordon TJ, Robergs RA. Prediction of one repetition maximum strength from multiple repetition maximum testing and anthropometry. J Strength Cond Res. 2006 Aug;20(3):584-92. doi: 10.1519/R-15304.1. PMID 16937972
- [Background] Nakayama A, Morita H, Nagayama M, Hoshina K, Uemura Y, Tomoike H, Komuro I. Cardiac Rehabilitation Protects Against the Expansion of Abdominal Aortic Aneurysm. J Am Heart Assoc. 2018 Feb 27;7(5):e007959. doi: 10.1161/JAHA.117.007959. PMID 29487112